CLINICAL TRIAL: NCT00387946
Title: An International, Seven-week, Double-blind, Placebo-controlled, Two Parallel Group Study to Assess the Efficacy of Dianicline 40 mg Bid as an Aid to Smoking Cessation in Cigarette Smokers
Brief Title: Efficacy and Safety of Dianicline Treatment as an Aid to Smoking Cessation in Cigarette Smokers (AMERIDIAN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5514; SSR591813
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Smoking Cessation; Tobacco Use Cessation
Keywords: smoking; cessation; tobacco
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation; Smoking | interventions — dianicline

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SSR591813L (dianicline)

SUMMARY:
The primary study objective is to demonstrate the efficacy of dianicline as an aid to smoking cessation in cigarette smokers. The main secondary objectives are to assess the: craving for cigarettes, nicotine withdrawal symptoms, and safety of dianicline.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, over legal age, smoking at least 10 cigarettes/day as a mean within the 2 months preceding the screening visit.

Exclusion Criteria:

* Patients who have taken an investigational drug within the past six months prior to the screening visit.
* Patients who had a previous quit attempt (= or >1 day with the aid of pharmacological adjunct) in the previous three months (before screening).
* Patients who have smoked or consumed non-tobacco cigarettes or any form of tobacco product (other than cigarettes such as cigars, pipes, smokeless tobacco, etc) more than 3 times within the 3 months preceding the screening visit.
* Patients who currently present with (based on Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition [DSM-IV]):

  * Psychotic disorder
  * Major depressive episode
* Pregnant or breast-feeding women.
* Women of childbearing potential not protected by effective contraceptive method of birth control and/or who are unwilling or unable to be tested for pregnancy. Medically acceptable methods of birth control for this study include approved hormonal contraceptive medications or devices, approved intra-uterine contraceptive devices, use of two combined barrier methods.
* Patients who have suffered from a myocardial infarction, unstable angina or other major cardiovascular event within the past week prior to screening.
* Patients who have a history of multiple allergic reactions to medications in two drug classes.
* Patients who have QTcF > 500 ms on the electrocardiogram (ECG).
* Patients with mild, moderate or severe renal impairment.
* Patients who have an abnormal laboratory test of potential clinical significance at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To assess the continuous abstinence from tobacco smoking at every visit during the last 4 weeks of treatment period, i.e. from week 4 to week 7, through direct inquiry of patients, exhaled carbon monoxide (CO) testing, and plasma cotinine measurements

SECONDARY OUTCOMES:
Questionnaire of Smoking Urges to assess craving for cigarettes; Hughes and Hatsukami Minnesota Withdrawal Scale to measure nicotine withdrawal, number of smoke-free days, and average number of cigarettes smoked from smoking status interview

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Administrative Office, Bridgewater, New Jersey, United States
- Administrative Office, Laval, Quebec, Canada

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273